CLINICAL TRIAL: NCT06266533
Title: Dismantling the U.S. Social Norm of the "Kids' Food" Archetype That Includes Ultra-processed Foods Such as Chicken Nuggets and Fries in the Newark, NJ Community
Brief Title: Dismantling the U.S. Social Norm of the "Kids' Food" Archetype (REACH Project)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Pamela Rothpletz-Puglia, EdD, RD, Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro2023002473
Record Dates: First submitted 2024-02-05; First posted 2024-02-20 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-04

CONDITIONS: Food Selection; Environmental Exposure
MeSH Terms: conditions — Food Preferences

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to a conventional nutrition education or an arts-based education group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Conventional Nutrition Education (Active Comparator): Conventional nutrition education
  Interventions: Behavioral: Conventional Ultra-processed Food Nutrition Education
- Arts-based Nutrition Education (Experimental): Arts-based nutrition education video production
  Interventions: Behavioral: Arts-based Ultra-processed Food Nutrition Education

INTERVENTIONS:
Behavioral: Conventional Ultra-processed Food Nutrition Education — The participants will receive a conventional nutrition education session with slides, flyers/handouts, and a lecture with discussion.
  Arms: Conventional Nutrition Education
Behavioral: Arts-based Ultra-processed Food Nutrition Education — The participants will receive an arts-based nutrition education session with video, animation, music, and discussion.
  Arms: Arts-based Nutrition Education

SUMMARY:
This project is the first stage of a health promotion campaign to shift social norms about marketing and feeding children ultra-processed foods. Embedded within a longitudinal ethnographic study using photo-elicitation techniques, mothers of preschool-age children will be randomly assigned to arts-based or traditional education about ultra-processed food.

DETAILED DESCRIPTION:
1. At baseline, describe how mothers of preschool-age children characterize food for children in their home and local environment and describe their knowledge of ultra-processed food.
2. To test different ways of providing nutrition education for increasing knowledge about children's nutrition and ultra-processed foods. Hypothesis: Both groups will correctly identify more ultra-processed foods post-education.
3. To learn in depth from mothers of preschool children about their perceptions of the food environmental culture (markets, advertising, health messaging, community norms, cultural norms, social norms) in Newark, NJ, through a series of focus group discussions about the mothers' photographs of the local food environment pre and post project.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* African American or Black or bi-racial or multi-racial African American and Black mothers
* >18 years
* Female
* Legal guardian of a preschool-age child (3-5 years) participating in the Leaguers, Inc.

Head Start programming.

Exclusion Criteria:

* Spanish-speaking
* Other racial and ethnic groups
* Fathers

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation
Enrollment: 38 (Actual)
Dates: Start 2024-02-21 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Ultra-Processed Food Knowledge | 60 minutes
  Participants will classify pictures of foods as ultra-processed or whole foods (adapted from Sarmiento-Santos, cited below) and as healthy or unhealthy. on a Pre and post-ultra-processed food knowledge questionnaire. Both sets of questions are yes or no categorical questions.
Environmental assessment of ultra-processed food | 6 months
  Participant photographs of the local food environment. At two time points (pre and post educational intervention) participants will take photographs of the local food environment including grocery stores, restaurant menus, etc. The purpose of this is to learn from participants about how they perceive the local kids' food environment and if they observe differences after the intervention. Photo elicitation techniques will be used during a series of focus groups for participants to discuss the photographs they took. These data will be analyzed using a layered analysis of the photographs (appraisal, discussion with participant who took the photo, cross-photo comparison, and interpretation) pre and post educational intervention, and thematic analysis of the focus group transcripts.

CONTACTS AND LOCATIONS:
Overall Officials: Pamela Rothpletz-Puglia, EdD, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- Leaguers Inc. Head Start, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sarmiento-Santos J, Souza MBN, Araujo LS, Pion JMV, Carvalho RA, Vanin FM. Consumers' Understanding of Ultra-Processed Foods. Foods. 2022 May 7;11(9):1359. doi: 10.3390/foods11091359. PMID 35564081
- [Background] Andreassen P, Christensen MK, Moller JE. Focused ethnography as an approach in medical education research. Med Educ. 2020 Apr;54(4):296-302. doi: 10.1111/medu.14045. Epub 2020 Feb 16. PMID 31850537
- [Background] Braun V, Clarke V. What can "thematic analysis" offer health and wellbeing researchers? Int J Qual Stud Health Well-being. 2014 Oct 16;9:26152. doi: 10.3402/qhw.v9.26152. eCollection 2014. No abstract available. PMID 25326092